CLINICAL TRIAL: NCT01831271
Title: Interventions for Patients With Cervical Radiculopathy- Neck-specific Training With a Cognitive Behavioural Approach Compared With Prescribed Physical Activity in a Prospective Randomised Controlled Trial
Brief Title: Neck-specific Training or Prescribed Physical Activity for Patients With Cervical Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Åsa Dedering, PhD, Head of Department, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KI: 2009/1756-31/4
Record Dates: First submitted 2013-04-05; First posted 2013-04-15 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Cervical Pain; Pain, Radiating
Keywords: Exercise, Physical; Physical Activity; Outcome Measures
MeSH Terms: conditions — Neck Pain; Pain; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prescribed physical activity (Other): Prescribed physical activity is a tailored physical activity programme with monitoring of progress and a follow-up. Also includes interview: exploratory talk, commitment/decision, life style change, health promotion, evaluation of readiness for change, reflection, assessment of motivation, patient specific goal assessment, conclusion and plan for follow-up at 14 weeks. Patients are guided by the physiotherapist to increase their overall activity and strength with i.e. walking and other self-mediated activities and exercise.
  Interventions: Other: Prescribed physical activity
- Neck specific training (Other): The active physiotherapy rehabilitation program consists of a standardised and structured physiotherapy program (twice a week) with medical exercise therapy and if needed vestibular rehabilitation. At the start of the intervention motivational interviewing will be included. Additionally once a week during the first 14 weeks of the program the physiotherapist informs the patient about physiology of pain, stress, exercise, breathing, relaxation, coping, pacing and ergonomics. All through the treatment program a cognitive approach from the physiotherapist according to theoretical behaviour change models will be used.
  Interventions: Other: Neck specific training

INTERVENTIONS:
Other: Prescribed physical activity — Prescribed physical activity is a tailored physical activity programme with monitoring of progress and a follow-up. Also includes interview: exploratory talk, commitment/decision, life style change, health promotion, evaluation of readiness for change, reflection, assessment of motivation, patient specific goal assessment, conclusion and plan for follow-up at 14 weeks. Patients are guided by the physiotherapist to increase their overall activity and strength with i.e. walking and other self-mediated activities and exercise.
  Arms: Prescribed physical activity
Other: Neck specific training — The active physiotherapy rehabilitation program consists of a standardised and structured physiotherapy program (twice a week) with medical exercise therapy and if needed vestibular rehabilitation. At the start of the intervention motivational interviewing will be included. Additionally once a week during the first 14 weeks of the program the physiotherapist informs the patient about physiology of pain, stress, exercise, breathing, relaxation, coping, pacing and ergonomics. All through the treatment program a cognitive approach from the physiotherapist according to theoretical behaviour change models will be used.
  Arms: Neck specific training

SUMMARY:
The overall objective is to evaluate if treatment with a neck-specific exercise program and cognitive behavioural approach improves the outcome compared with prescribed, self-mediated and progressive physical activity in patients with cervical radiculopathy. There is a lack of evidence of the best treatment for the patient category. Many patients are sick-listed for long periods of time with different kind of treatment approaches or without any treatment at all. The present study could fill the identified knowledge gap by strengthening of the currently weak scientific evidence for treatment of the patient category. The long-term effects of the study could be to reduce the time for sick leave and improve the rate of patients returning to work and/ or former activity by optimising treatments. Further on, to decrease the number of patients who finally have surgery for their neck problems and thus reducing the mental, physical and social costs.

DETAILED DESCRIPTION:
Patients with cervical radiculopathy have neck- and arm pain, neurological changes, activity limitations and difficulties in returning to work. The current scientific evidence lacks randomised controlled trials to compare surgery with conservative treatment as well as to evaluate different conservative interventions. Most patients are not candidates for surgery and are sick-listed for long time with different treatment approaches or without any treatment at all. The purpose is to evaluate if treatment with neck-specific training and a cognitive behavioral approach improves the outcome compared with prescribed physical activity. Methods: A randomized controlled trial including 144 patients will compare the intervention neck specific training and cognitive behavioural approach with an intervention of prescribed physical activity. The interventions will be led by experienced and specialised physiotherapists and last 14 weeks. Main outcome variable is pain intensity (VAS scale) accompanied with assessments of impairments and subjective health measurements undertaken before intervention and at 3, 6, 12 and 24 months. Implementation: The results will be presented scientifically as well as popularly in publications and professional meetings. Active implementation strategies to change physiotherapists treatment behaviour will be used. The best method will be chosen after surveying the physiotherapists treating patients in the current study regarding experiences, education and organisational context.

ELIGIBILITY:
Inclusion Criteria:

* Magnetic Resonance Imaging (MRI) verified cervical disc disease showing cervical nerve root compression
* Positive Spurling sign and/or cervical extension test
* Clinical examination signs matching the MRI

Exclusion Criteria:

* earlier fracture or luxation of the cervical column,
* malignity,
* spinal tumour,
* spinal infection,
* previous surgery in the cervical column,
* co-morbidity such as disease or symptoms contraindicated to perform the treatment program or the measurements,
* known drug abuse,
* lack of familiarity with the Swedish language,
* diagnosed psychiatric disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2010-08; Primary Completion 2016-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Pain | Baseline and change after 15 weeks, 6 months, 1 year, 2 years follow up. The outcome measures is going to report a change over time.
  Neck and Arm Pain is measured with Visual Analogue Scale

SECONDARY OUTCOMES:
Disability | Baseline and change after 15 weeks, 6 months, 1 year, 2 years follow up. The outcome measures is going to report a change over time.
  Neck Specific Disability is measured with Neck Disability Index (NDI)

OTHER OUTCOMES:
Health related quality of life | Baseline and change after 15 weeks, 6 months, 1 year, 2 years follow up. The outcome measures is going to report a change over time.
  Health related quality of life is assessed by the EuroQuol 5 dimensions (EQ-5D).
Self-efficacy | Baseline and change after 15 weeks, 6 months, 1 year, 2 years follow up. The outcome measures is going to report a change over time.
  Self-efficacy will be measured on the Self-efficacy and Exercise Self-efficacy scales
Symptom satisfaction | Baseline and change after 15 weeks, 6 months, 1 year, 2 years follow up. The outcome measures is going to report a change over time.
  Symptom satisfaction is rated on 7-grade scale
Fear Avoidance Beliefs | Baseline and change after 15 weeks, 6 months, 1 year, 2 years follow up. The outcome measures is going to report a change over time.
  Fear Avoidance Beliefs will be measured with Fear Avoidance Beliefs questionnaire (FABQ)and Tampa scale (TSK)
Depression | Baseline and change after 15 weeks, 6 months, 1 year, 2 years follow up. The outcome measures is going to report a change over time.
  Hostility, anxiety and depression will be measured with Hostility, anxiety and depression scale (HAD)
Coping strategies | Baseline and change after 15 weeks, 6 months, 1 year, 2 years follow up. The outcome measures is going to report a change over time.
  Coping strategies will be measured with Coping strategy questionnaire
Pain catastrophizing | Baseline and change after 15 weeks, 6 months, 1 year, 2 years follow up. The outcome measures is going to report a change over time.
  Pain catastrophizing will be measured with Pain catastrophizing scale
Physical activity | Baseline and change after 15 weeks, 6 months, 1 year, 2 years follow up. The outcome measures is going to report a change over time.
  Physical activity will be measured with International Physical activity questionnaire
Patients specific goals | Baseline and change after 15 weeks, 6 months, 1 year, 2 years follow up. The outcome measures is going to report a change over time.
  Patients specific goals will measured with Patients specific functional scale and Patient goal assessment scale
Work ability | Baseline and change after 15 weeks, 6 months, 1 year, 2 years follow up. The outcome measures is going to report a change over time.
  Work ability will be measured with Work Ability Index
Physical clinical outcome measures | Baseline and change after 15 weeks, 6 months, 1 year, 2 years follow up. The outcome measures is going to report a change over time.
  Clinical examination
Cervical range of motion | Baseline and change after 15 weeks, 6 months, 1 year, 2 years follow up. The outcome measures is going to report a change over time.
Hand strength | Baseline and change after 15 weeks, 6 months, 1 year, 2 years follow up. The outcome measures is going to report a change over time.
Muscle fatigue | Baseline and change after 15 weeks, 1 year follow up. The outcome measures is going to report a change over time.
  Electromyography on the neck muscles
Neck muscle endurance | Base line, 15 weeks, 6 months, 1 year, 2 years, The outcome measures is going to report a change over time.
  Neck muscle endurance time measured in sec for dorsal and ventral neck muscles during a static endurance test

CONTACTS AND LOCATIONS:
Overall Officials: Åsa Dedering, PhD, Study Chair — Karolinska Institutet
Locations (1):
- Department of Physical Therapy, Karolinska University Hospital,, Stockholm, Sweden

REFERENCES:
- [Background] Dedering A, Halvorsen M, Cleland J, Svensson M, Peolsson A. Neck-specific training with a cognitive behavioural approach compared with prescribed physical activity in patients with cervical radiculopathy: a protocol of a prospective randomised clinical trial. BMC Musculoskelet Disord. 2014 Aug 12;15:274. doi: 10.1186/1471-2474-15-274. PMID 25115308
- [Derived] Dedering A, Peolsson A, Cleland JA, Halvorsen M, Svensson MA, Kierkegaard M. The Effects of Neck-Specific Training Versus Prescribed Physical Activity on Pain and Disability in Patients With Cervical Radiculopathy: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2018 Dec;99(12):2447-2456. doi: 10.1016/j.apmr.2018.06.008. Epub 2018 Jul 4. PMID 30473018